CLINICAL TRIAL: NCT00382525
Title: Phase IV Long Term Observational Study of Patients Implanted With Medtronic CRDM Implantable Cardiac Devices
Brief Title: PANORAMA Observational Study
Status: Completed | Type: Observational
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Other Study IDs: Version 1 April 25th, 2005
Record Dates: First submitted 2006-09-28; First posted 2006-09-29 (Estimated); Last update posted 2025-07-03 (Actual); Status verified 2017-09

CONDITIONS: Arrhythmia; Sinus Node Disease; Heart Failure; Heart Block
Keywords: Bradyarrhythmia; Atrial Fibrillation; Ventricular Tachycardia; Ventricular Fibrillation; Heart Failure; Pacemaker; Implantable Cardioverter Defibrillator; Cardiac Resynchronization Therapy; Loop recorder; Registry
MeSH Terms: conditions — Arrhythmias, Cardiac; Sick Sinus Syndrome; Heart Failure; Heart Block; Bradycardia; Atrial Fibrillation; Tachycardia, Ventricular; Ventricular Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with Cardiac Rhythm Management device: Patients receiving a Medtronic Cardiac Rhythm Device, worldwide
  Interventions: Device: Cardiac Rhythm Management device

INTERVENTIONS:
Device: Cardiac Rhythm Management device

SUMMARY:
To construct a computerized database of national profiles and epidemiological data on patients wearing Medtronic implantable pacemakers and cardioverter defibrillators (both with or without cardiac resynchronization therapy), implantable loop recorders and leads used within their intended use.

Clinical variables will be analyzed in relation to device-based data and diagnostics.

DETAILED DESCRIPTION:
PANORAMA will collect a large database of device behavior, for instance to monitor long term behavior of device features, technical reliability and longevity, as well as to allow studying device performance in different subgroups of patients. Larger databases are often essential for formulating and testing study hypotheses for prospective (randomized) trials. While it may depend on specific objectives for individual devices, reliable assessment of device performance over longer periods and in broad patient populations typically requires a study population from a few hundred to a few thousand patients. PANORAMA collects acute and chronic patient and device data in a large population during routine usage of the device, without specific study interventions, and always within the approved intended use of the device.

In the past, observational studies were designed and conducted specifically on a device-by-device case. PANORAMA avoids the redesign of the same set of data. It establishes a core database which can be expanded with substudies creating more detailed data sets for particular CRDM devices/features.

PANORAMA will be open for inclusion to any patient (to be) implanted with a CRDM device. It shall be suitable for current and upcoming CRDM devices implanted in patients. It will serve as an epidemiological tool designed to stratify morbidity and mortality of all cardiac diseases treated by implantable CRDM devices.

ELIGIBILITY:
Inclusion Criteria:

* (To be) implanted with a Medtronic market-released cardiac device,
* Signed Patient Data Release Form.

Exclusion Criteria:

* Unwillingness or inability to cooperate or give voluntary consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients receiving market released Medtronic Cardiac Rhythm device, worldwide
Sampling Method: Non-Probability Sample
Enrollment: 8586 (Actual)
Dates: Start 2005-01; Primary Completion 2012-10 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
To construct a computerized database of national profiles and epidemiological data on patients wearing Medtronic Cardiac Rhythm Management Devices | 2013
  To construct a computerized database of national profiles and epidemiological data on patients wearing Medtronic implantable pulse generators [IPG] and implantable cardioverter defibrillators [ICD] both with or without cardiac resynchronization therapy [+/- CRT], implantable loop recorders [ILR] and leads implanted within intended use.
  Stratified per country, per pathology, per indication and per device type.

CONTACTS AND LOCATIONS:
Locations (27):
- Belgium (6):
  - C.H.I.R.E.C. - Site de Braine la Alleud, Braine-l'Alleud
  - A.Z. Klina, Brasschaat
  - St. Vincentius-Campus St. Jozef, Mortsel
  - Centre de Medecine Cardiologique, Namur
  - Centre Hosp. Régional du Tournaisis- Site Hopital, Tournai
  - Hôpital Notre Dame de Tournai, Tournai
- India (2):
  - S.A.L. Hospital and Medical Institute, Ahmedabad
  - Max Devki Devi Foundation, New Delhi
- Chest Disease Hospital, Safat, Kuwait
- Russia (14):
  - Regional Clinical Cardio Center, Khabarovsk
  - FGU Moscow SRC of Pediatrics & Childrens Surgery, Moscow
  - Scientific Center of Heart Surgery by A.N. Bakulev, Moscow
  - Scientific Research Institute of Transplantology, Moscow
  - Novosibirsk Regional Cardio Center, Novosibirsk
  - Scientific Research Institute of Circ. Pathology, Novosibirsk
  - Rostov area hospital, Rostov-on-Don
  - I.P. Pavlovs State Medical University- Hospital #2, Saint Petersburg
  - Medical Academy of Postgraduate Studies, Saint Petersburg
  - Scientific Research Insitute of Cardiology, Tomsk
  - Tyumen Cardiology Center, Tyumen
  - Regional Hospital #1, Vladivostok
  - Volgograd cardio center, Volgograd
  - Sverlovsk Regional Clinical Hospital N1, Yekaterinburg
- Sweidan Raed King Fahd Armed Forces Hospital, Jeddah, Saudi Arabia
- Serbia and Montenegro (3):
  - Cardiovascular Institute Dedinje, Beograd (Belgrade)
  - Clinical Centre Nis, Nis
  - Instit. of Cardiovasc. Diseases, Univ. of Novi Sad, Sremska Kamenica